CLINICAL TRIAL: NCT06083623
Title: A Randomized, Double-blind, Placebo-controlled and Parallel Group Adaptive Phase 2b/3 Trial to Evaluate the Efficacy and Safety of TNM001 Injection for the Prevention of Lower Respiratory Tract Infection Caused by Respiratory Syncytial Virus in Infants Under One Year of Age
Brief Title: A Trial to Evaluate the Efficacy and Safety of TNM001 for the Prevention of Lower Respiratory Tract Infection Caused by Respiratory Syncytial Virus in Infants
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TNM001-301; CTR20232792 (Other: ENTER FOR DRUG EVALUATION, NMPA)
Record Dates: First submitted 2023-09-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNM001 (Experimental)
  Interventions: Biological: TNM001
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: TNM001 — single dose intramuscular injection
  Arms: TNM001
Biological: placebo — single dose intramuscular injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, pharmacokinetics (PK), neutralizing antibody and antidrug antibody (ADA) response for TNM001 in infants entering their first RSV season.

DETAILED DESCRIPTION:
This study adopts an adaptive seamless dose selection design and consists of two parts: Part 1 is a phase 2b dose ranging trial which will support to determine the dose for Part 2, the phase 3 trial. The study population includes early and mid-term preterm infants [gestational age (GA)﹤35 weeks 0 day] and late preterm infants or full-term infants (≥35 weeks 0 day GA), with or without Congenital Heart Disease (CHD) or premature infants Chronic Lung Disease (CLD). A total of approximately 2250 infants will be randomized 2:1 to receive either TNM001 or placebo. All subjects will be followed for 240 days after dosing. This study will be conducted in appropriately 50 sites in China.

ELIGIBILITY:
Inclusion Criteria:

* 1. Early and mid-term preterm infants (<35 weeks 0 day GA) and late preterm infants or full-term infants (≥35 weeks 0 day GA) under 1 year of age, with or without Congenital Heart Disease (CHD) or premature infants Chronic Lung Disease (CLD)，who are entering their first RSV season at the time of screening.

Exclusion Criteria:

* 1. Any fever (> 38.0°C) or acute illness within 7 days prior to randomization
* 2. History of RSV infection or active RSV infection prior to, or at the time of, randomization
* 3. Drug medication prior to randomization or expected to be treated by medicines during the study period.
* 4. Currently receiving or expected to receive immunosuppressive therapy during the study period.
* 5. Renal impairment or hepatic dysfunction
* 6. Nervous system disease or neuromuscular disease
* 7. Prior history of a suspected or actual acute life-threatening event
* 8. Known immunodeficiency including HIV, mother with HIV infection unless the child's infection has been excluded.
* 9. Known allergy history of immunoglobulin products, receipt or expected to receive immunoglobulins or blood products during the study period.
* 10.Receipt of RSV vaccine or mAb

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2250 (Estimated)
Dates: Start 2023-10-06 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of medically attended LRTI due to RT-PCR confirmed RSV | 150 days post dose

SECONDARY OUTCOMES:
Incidence of hospitalization due to RT-PCR confirmed RSV LRTI | 150 days post dose
Occurrence of adverse events (AEs) | 240 days post dose
Change in body temperature (celsius) | 240 days post dose
Change in blood pressure (mmHg) | 240 days post dose
Change in heart rate (beats per minute) | 240 days post dose
Change in respiratory rate (breaths per min) | 240 days post dose
Number of subjects with clinical significant abnormality in physical examinations | 240 days post dose
Serum concentration of single dose TNM001 at pre-specified timepoints | 240 days post dose
Serum level of neutralizing antibody to RSV | 240 days post dose
Positive rate of anti-drug antibody (ADA) to TNM001 in serum | 240 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Hanmin Liu, MD, Principal Investigator — West China Second Hospital, Sichuan University; Enmei Liu, MD, Principal Investigator — Children's Hospital of Chongqing Medical University; Ying Wang, Study Director — Zhuhai Trinomab Pharmaceutical Co., Ltd.
Locations (39):
- China (39):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Children's Hospital Capital Institute Pediatrics, Beijing, Beijing Municipality
  - Jiangjin Central Hospital, Chongqing, Chongqing Municipality
  - Xiamen maternal and Child Health Hospital, Xiamen, Fujian
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangdong, Guangdong
  - Guangdong Maternal and Child Health Care Hospital, Guangzhou, Guangdong
  - University of Chinese Academy of Sciense Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - LiuZhou People's Hospital, Liuchow, Guangxi
  - Maternity and Child Health Care of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - HaiNan Women and Children's Medical Center, Haikou, Hainan
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of HeBei Medical University (HBMU), Shijiazhuang, Hebei
  - Tangshan Maternal and Child Health Hospitaltangshan Maternal and Child Health Hospital, Tangshan, Hebei
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Xinxiang First People's Hospital, Xinxiang, Henan
  - Henan (Zhengzhou) Children's Hospital, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - The First People'S Hospital of Changde City, Changde, Hunan
  - The Maternal and Child Health Hospital of Hunan Province, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Hospital University of South China, Hengyang, Hunan
  - Loudi Central Hospital, Loudi, Hunan
  - The First Affiliated Hospital of Shaoyang University, Shaoyang, Hunan
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Children's Hospital Affiliated to Shandong University, Jinan, Shandong
  - The affiliated children'shospital fudan university, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Children's Hospital of Chongqing Medical University, Chongqing, Sichuan
  - Mianyang Peoples Hospital, Mianyang, Sichuan
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine/Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Ningbo Women&Children's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided